CLINICAL TRIAL: NCT01297959
Title: Phase 3 Study of Efficacy and Safety of Topical E-101 Solution to Prevent Incisional Infections Among Colorectal Surgery Patients (Triple IN Study --Inhibition of Incisional Infections)
Brief Title: Study to Evaluate Efficacy and Safety of E-101 Solution for Preventing Surgical Site Infections After Colorectal Surgery
Acronym: Triple IN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Excited States, LLC (Industry)
Collaborators: Veristat, Inc. (Other); Biotec Services International Ltd (Other); Eurofins (Industry); CBR International Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E-101:PH3:2012:004
Record Dates: First submitted 2011-02-11; First posted 2011-02-17 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Infections
Keywords: Surgical Wound Infection; Therapeutic Enzyme System; Singlet Oxygen; Peroxidase; Glucose Oxidase; Colorectal surgery; Incisional Surgical Site Infections (SSI); Anti-infective Agents, Local; Clinical Trial, Phase III
MeSH Terms: conditions — Infections; Surgical Wound Infection | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E-101 Solution 300 GU/mL (Experimental): Participants will receive E-101 Solution at porcine myeloperoxidase (pMPO) concentration of 300 guaiacol units per milliliter (GU/mL) applied topically twice to surgical wound site. The first topical application will occur just after incision to the level of the rectus fascia or linea alba without penetration through the peritoneum and the second topical application will occur just after closure of the rectus fascia or linea alba but prior to closure of the incisional wound.
  Interventions: Drug: E-101 Solution 300 GU/ml
- Placebo (Saline solution) (Placebo Comparator): Participants will receive placebo (saline solution) matched to E-101 Solution applied topically twice to surgical wound site. The first topical application will occur just after incision to the level of the rectus fascia or linea alba without penetration through the peritoneum and the second topical application will occur just after closure of the rectus fascia or linea alba but prior to closure of the incisional wound.
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: E-101 Solution 300 GU/ml — 8 mL of E-101 Solution
  Arms: E-101 Solution 300 GU/mL
Drug: Saline solution — Saline solution matched to E-101
  Arms: Placebo (Saline solution)

SUMMARY:
This study is intended to determine the efficacy, safety and tolerability of topical application of E-101 Solution directly into the surgical incisional wound in the prevention of infection of superficial and deep surgical incisional wounds. E-101 Solution is an enzyme-based antiseptic that is being developed for direct application to a surgical incision.

DETAILED DESCRIPTION:
The purpose of this standard-of-care, pivotal Phase 3 study is to evaluate the efficacy and safety of topical E-101 Solution after direct application into the principal surgical incision in the prevention of superficial and deep incisional surgical site infections (SSI) within 30 days after elective colorectal surgery. The study is intended to support a target indication statement of: "E-101 Solution is indicated for the prophylaxis of incisional surgical site infections following elective colorectal surgery". E-101 Solution is comprised of the active ingredients of glucose oxidase (GO) and porcine myeloperoxidase (pMPO) that produce coupled reactions after the addition of glucose substrate. The hypothesis is that E-101 Solution topically applied directly into the principal incision is safe and significantly reduces the incidence of incisional SSI compared to placebo topical application. (The principal surgical incision is ≥ 5cm and < 35 cm used as a hand port, colorectal specimen extraction port, or extracorporeal manipulation port depending on the specific colorectal surgical approach.)

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo elective colon and/or rectal surgical procedures involving open laparotomy, hand-assisted laparoscopy, and laparoscopic-assisted approaches. The principal incision must have a length of > 5 cm and < 35 cm in length. Eligible surgeries are: left hemicolectomy, right hemicolectomy, transverse colectomy, ileocolic resection, total abdominal colectomy with ileorectal anastomosis, total abdominal proctocolectomy (portion of specimen to be extracted via laparotomy), low anterior resection, sigmoid resection, non-emergent Hartmann procedure, colostomy takedown through laparotomy (not peristomal) incision, ileo-pouch anal anastomosis, and abdominal perineal resection of the rectum.
2. Able to give informed consent.
3. If female, is non-pregnant (negative pregnancy test result at the Screening/Randomization Visit) and non-lactating.
4. If female, is either not of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [status post bilateral tubal occlusion, bilateral oophorectomy, or hysterectomy]) or practicing 1 of the following methods of birth control and agrees to continue with this regimen over the study surveillance period:

   * Oral, implantable, or injectable contraceptives for 3 consecutive months before the Baseline/Randomization Visit
   * Intrauterine device
   * Double barrier method (condoms, sponge, or diaphragm with spermicidal jellies or cream)
   * Not sexually-active. Agreement to be available for evaluation at the study site for scheduled visits.

Exclusion Criteria:

1. Hypersensitivity to porcine products.
2. History of known anti-myeloperoxidase autoantibodies (i.e., perinuclear anti-neutrophil cytoplasmic antibody [pANCA]), as well as participants with known idiopathic necrotizing glomerulonephritis and certain systemic vasculitis conditions [e.g., microscopic polyangiitis of small blood vessels, Wegener's granulomatosis, and Churg-Strauss Syndrome]).
3. Use of microbial sealant (IntegusealTM), any antibiotic-embedded suture, or any antimicrobial-embedded suture to close the principal incision or any suture in the surgical field that has not been formally approved by the relevant local national regulatory authority.
4. Absolute contraindication to general anesthesia.
5. Hypersensitivity reactions to steri-strip tapes, medical-surgery tapes, adhesives, or sutures. (Note: If there can be assurances that the participant will not be exposed to these materials that cause hypersensitivity, alternatives will be allowed.)
6. History of keloid or hypertrophic scarring within or near an incision from a prior surgery.
7. Body mass index [BMI]: > 50 or < 20 (both due to the extremely high risk of poor wound healing).
8. American Society of Anesthesiologists (ASA) Score > 3.
9. Undergoing emergency colorectal surgery such that standard bowel preparation and other standard preoperative precautions and assessments cannot be performed in time before the index-surgery.
10. The planned index-surgery involves removal or placement of mesh (either synthetic or biological) as part of closure in the principal incision or traversing any part of a pre-existing mesh (either synthetic or biological) in the principal incision.
11. There are clinical signs of overt infection necessitating systemic antibiotics via oral, intramuscular, or intravenous routes (e.g., infection of the abdominal wall, peritonitis, pneumonia, and sepsis/septic shock) prior to the index-surgery.
12. Preoperative severe neutropenia (total neutrophil count ≤500 X 109/L). (Note: Testing should be performed at the local laboratory.)
13. Receiving any oral or intravenous antibiotics within 24 hours prior to the index-surgery. (Note: It is permissible to administer conventional oral prophylactic antibiotics as bowel preparation up to the time of the index- surgical procedure, as well as intravenous or intramuscular prophylactic antibiotics just prior to the index-surgery as per the treating surgeon's standard of care.)
14. Preoperative evaluation that the intra-abdominal process might preclude full closure of the skin incision due to severe or morbid obesity (i.e., any mechanical reason that would prevent/preclude primary intent wound healing) at the principal incision.
15. History of major organ transplantation (e.g., lung, liver, or kidney), including bone marrow transplantation, or intent to perform major organ transplant as a concomitant surgery.
16. History of a complicated laparotomy within 30 days prior to planned index-surgery.
17. Planning to undergo a second colorectal surgical procedure (e.g., colostomy or ileostomy takedown) or any other general surgery in less than 30 days of index-surgery.
18. Likely preoperative urinary tract infection, as evident by: i) symptoms of upper urinary tract infection (e.g., fever and/or flank pain) or ii) symptoms of lower urinary tract infection (e.g., urinary frequency, dysuria, urgency, and/or suprapubic pain); accompanied by any one of the following: 1) bacteriuria of ≥104 bacteria/mL urine or 2) positive urine leucocyte esterase or positive nitrite urine dipstick tests. Also exclude any man under age 60 years who has both positive urine nitrite and leucocyte esterase dipstick tests - even if he is asymptomatic (unless he has predisposing factors for urinary tract infection - e.g., spinal cord injury). (Note: Testing should be performed at the local laboratory.)
19. Undergoing a significant concomitant surgical procedure (e.g., hysterectomy) or any mesh repair (either synthetic or biological mesh) as part of closure. The following concomitant procedures are allowed: appendectomy, cholecystectomy, oophorectomy, removal of Meckel's diverticulum, primary repair of small ventral hernia (i.e., <30 cm2), liver biopsy/wedge resection (but not liver resection).
20. Participants with a condition (e.g., recurrent urinary tract infections, nail infections, sinusitis, dental infections, vaginitis/vaginosis, or chronic bronchitis) requiring frequent or chronic administration of antimicrobials (received antibiotics/antimicrobials at least twice for ≥ 2 weeks during past 6 months).
21. Preoperative prothrombin time or international normalized ratio (INR) > 2 x upper limit of normal. (Note: Testing should be performed at the local laboratory.)
22. Postsurgical life expectancy ≤ 60 days (in the Investigator's or Sponsor's opinion).
23. Any participant in which the planned surgery would include: i) placement of a stoma in the principal incision; ii) placement of a drain into the supra-peritoneal fascia space that emerges through the principal incision; iii) placement of a drain into the intraperitoneal space that emerges through the principal incision; and iv) supplementation of any of the irrigation fluid with antibiotic or antiseptic drugs.
24. Participant with severe Chronic obstructive pulmonary disease (COPD) that are likely to need > 24 hours postoperative ventilator support (e.g. participant on chronic or intermittent supplemental oxygen or an estimated forced expiratory volume in 1 second (FEV1) less than 50% of expected based on bedside spirometry).
25. If, in the opinion of Investigator, the potential participant would likely be unable to maintain adequate care of the principal incision post-operatively.
26. Anticipate that participant will not be available for study visits/ procedures or if in the opinion of Investigator there is concern that participant might not comply with study visits/procedures (e.g., due to ongoing illicit drug usage or alcohol abuse).
27. Lack of willingness to have personal study-related data collected, archived, or transmitted under a blinded condition to regulatory agencies.
28. Participation within 30 days before the start of this study in any experimental drug or device study; or currently participating in a study in which the administration of investigational drug or device within 60 days is anticipated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2015-10-14 (Actual); Study Completion 2015-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Hanley, PhD, MD, MPH, Study Director — Excited States, LLC; Robert Martindale, MD, PhD, Study Chair — Oregon Health and Science University; Michael J Stamos, MD, Principal Investigator — University of California, Irvine; Jerrold H Levy, MD, Principal Investigator — Emory Healthcare
Locations (39):
- United States (34):
  - University of South Alabama Medical Center, Mobile, Alabama
  - University of Southern California, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Sheridan Clinical Research, Inc., Sunrise, Florida
  - University of South Florida/Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Stoger Hospital of Cook County, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Colon & Rectal Surgery Associates, Metairie, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation / Colon and Rectal Surgery, New Orleans, Louisiana
  - Berkshire Medical Center, Inc, Pittsfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Medical IQ, Brandon, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Colon and Rectal Surgery, Inc., Omaha, Nebraska
  - CentraState Medical Center, Freehold, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Meridian Health Jersey Shore University Medical Center, Neptune City, New Jersey
  - Albany Medical Center, Albany, New York
  - Mount Sinai School of Medicine, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Baylor Research Institute, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Southwest Surgical Associates, L.L.P., Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Southwest Surgical Associates, LLP, Sugar Land, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadasit Medical Research Services & Development LTD, Jerusalem
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky

REFERENCES:
- [Result] Denys, G.A., O'Hanley P, Stephens, JT. E-101 Solution demonstrates antiviral properties against Herpes Simplex Virus, Human Immunodeficiency Virus, and Human Influenza A/H1N1 Virus. American Society for Microbiology, 110th General meeting, San Diego, CA (Abstract # C-2061). May 2010.
- [Result] O'Hanley, P, Beausoleil C, O'Hanley K, Stephens, JT. E-101 Solution, a novel antiseptic intended for direct application within a surgical wound to prevent surgical site infection: Blinded, controlled Phase 1 skin irritation study in healthy volunteers. Annual Surgical Site Infection Meeting, Las Vegas, NV, May 2010.
- [Result] O'Hanley P, O'Hanley K, Beausoleil C, Stephens JT. E-101 Solution (E-101), a Myeloperoxidase (MPO) Antiseptic for Prevention of Surgical Site Infections (SSI): Phase 1 Sensitization and Microbial Reduction in Healthy Adult Volunteers. Program and Abstracts of the 50th Interscience Conference on Antimicrobial Agents and Chemotherapy, Boston, MA, October 2010.
- [Result] Pillar, C, Denys GA, O'Hanley P, Stephens JT, Sahm D. E-101, a novel in class topical anti-infective, has potent activity against clinical isolates of important pathogens in Europe collected from 2008-2010. 21st ECCMID/27th ICC, Milan, Italy, May 2011.
- [Result] Pillar C, Denys GA, O'Hanley P, Stephens JT, Sahm D. E-101, a novel in class topical anti-infective, maintains a high degree of potency in vitro against problematic resistant clinical pathogens (ESKAPE pathogens). 21st ECCMID/27th ICC, Milan, Italy, May 2011.
- [Result] Denys, GA, Goheen MP, Allen RC, O'Hanley P, Stephens JT. Effect of E-101 Solution and its oxidative products on microbial ultrastucture changes associated with microbicidal action. 21st ECCMID/27th ICC, Milan, Italy, May 2011.
- [Result] O'Hanley, P, Pete M, O'Hanley K, Sabo L, Allen R, Stephens JT. Antibody Responses Not Likely to Affect Efficacy and Safety of E-101 Solution, a Novel Myeloperoxidase (MPO)-based Topical Antiseptic for Prevention of Incisional Infections. Annual Surgical Site Infection Society Meeting, Palm Beach, FL, May 2011.
- [Result] Denys GA, Allen RC, O'Hanley P, Stephens JT. E-101 solution, a first in class topical anti- infective, shows fungicidal activity in vitro against Candida species. 11th ASM Conference on Candida and Candidiasis March 29-April 2, 2012 San Francisco, CA.
- [Result] Deane J, Simenauer A, Denys GA, O'Hanley P, Stephens JT, Sahm DF. In vitro activity of E-101, a rapidly bactericidal myeloperoxidase (MPO)-based agent, against key bacterial pathogens. 52nd Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC), September 9-12, 2012 San Francisco, CA.
- [Result] Denys GA, Shah D, Deane D, Sahm DF, O'Hanley P, Stephens JT. Antimicrobial susceptibility of E-101 Solution against target aerobic pathogens: A 5-year longititudional study. 53rd Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC), September 9-13, 2013 Denver, CO.
- [Result] Denys, GA, MP Goheen, RC Allen, P O'Hanley, JT Stephens Jr. Antifungal activity of two potent topical haloperoxidase-based formulations (EPO-based C-101 and MPO-based E- 101) against Candida albicans. American Society for Microbiology, 114th General Meeting, Boston MA (Abstract #681). May 17-20, 2014.
- [Result] Denys, GA, C Schneider, P O'Hanley, JT Stephens, Jr., K Babcock. Use of Affinity Biosensor's LifeScale resonant mass measurement to assess antimicrobial activity of E-101 solution, a novel haloperoxidase-based topical antimicrobial agent. American Society for Microbiology, Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC), Washington, DC (Abstract F-1573). September 5-9, 2014.
- [Result] Denys, GA, KM Koch, RC Allen, P O'Hanley, JT Stephens, Jr. Superiority of E- 101 solution, a haloperoxidase-containing enzyme product, to sodium oxychlorosene as an antiseptic agent in the presence of serum and whole blood. American Society for Microbiology, 115th General Meeting, New Orleans, LA. May 30-June 2, 2015.
- [Result] Denys GA, Shah D, Sahm DF, Allen RC, O'Hanley P. Stephens JT. In vitro activity of C- 101 solution, a new eosinophil peroxidase (EPO) containing enzyme system, against Gram- negative and Gram-positive pathogens. 52nd Interscience Conference on Antimicrobial Agents and Chemotherapy (ICAAC), September 9-12, 2012 San Francisco, CA.

RESULTS

PARTICIPANT FLOW:
Groups:
- E-101 Solution 300 GU/mL: Participants received 8 milliliter (mL) of E-101 Solution at porcine myeloperoxidase (pMPO) concentration of 300 guaiacol units per milliliter (GU/mL) applied topically twice to surgical wound site. The first topical application occurred just after incision to the level of the rectus fascia or linea alba without penetration through the peritoneum and the second topical application occurred just after closure of the rectus fascia or linea alba but prior to closure of the incisional wound.
- Placebo (Saline Solution): Participants received placebo (saline solution) matched to E-101 Solution applied topically twice to surgical wound site. The first topical application occurred just after incision to the level of the rectus fascia or linea alba without penetration through the peritoneum and the second topical application occurred just after closure of the rectus fascia or linea alba but prior to closure of the incisional wound.
Period: Overall Study
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Started | 261 | 242
Completed | 241 | 226
Not Completed | 20 | 16
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Unrelated medical illness / complication | 0 | 2
Not completed — Other | 13 | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomized to treatment and exposed to any quantity of study drug.
Groups:
- E-101 Solution 300 GU/mL: Participants received 8 mL of E-101 Solution at pMPO concentration of 300 GU/mL applied topically twice to surgical wound site. The first topical application occurred just after incision to the level of the rectus fascia or linea alba without penetration through the peritoneum and the second topical application occurred just after closure of the rectus fascia or linea alba but prior to closure of the incisional wound.
- Total: Total of all reporting groups
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution) | Total
Number analyzed (Participants) | 248 | 234 | 482
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (14.68) | 59.7 (14.36) | 59.7 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 93 | 200
  Male | 141 | 141 | 282
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 5 | 4 | 9
  Race: Black | 28 | 19 | 47
  Race: White | 211 | 208 | 419
  Race: Others | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 8 | 7 | 15
  Ethnicity: Not Hispanic or Latino | 235 | 225 | 460
  Ethnicity: Not Reported | 3 | 1 | 4
  Ethnicity: Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants In Intent to Treat (ITT) Analysis Set With Superficial and Deep Incisional Surgical Site Infections (SSI) Involving Principal Incision Within 30 Days After Index-surgery as Determined by Blinded Assessors 30 Days Post-operatively
Description: Superficial SSI: purulent drainage (PD) from superficial incision (SI), organisms isolated from aseptically obtained culture fluid from SI, pain/tenderness, localized swelling, redness, or heat extending from principal incision (PI), or PI deliberately opened by surgeon for presumptive PI infection and was culture-positive, a negative wound culture but clinical evidence of infection on Clinical Infection Wound Scale (CIWS). Deep incisional SSI: PD from deep incision (DI) but not from organ/space component of the surgical site, fever (>38°C), localized wound pain, or wound tenderness, or DI spontaneously dehisces and/or deliberately opened by surgeon, and microbiological culture of DI by aseptic collection or deep wound swab was positive, an abscess or other evidence of infection involving DI was found on direct examination, during reoperation, or by histopathological or radiological examination, negative deep wound culture but clinical evidence of deep wound infection on CIWS.
Time Frame: Surgery (Day 0) up to 30 days post-surgery
Population: ITT Analysis Set included all randomized participants in their assigned treatment group except those were found between randomization and before surgery to either meet exclusion criteria or not meet inclusion criteria, who withdrew consent or were treated at site 03-03 (participants were excluded because of a systematic problem in incisional SSI surveillance due to a lack of blinded assessors). Cumulative Treatment Incisional SSI was reported which included Superficial SSI and Deep SSI.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 241 | 225
Participants | 53 | 41
Statistical Analysis 1: Comparison: E-101 Solution 300 GU/mL vs Placebo (Saline Solution); Test type: Superiority; p = 0.39, Regression, Logistic; p-value was based on a logistic regression (Chi-square test) model with treatment group as a factor, adjusting for the stratification factors

2. Primary Outcome: Number of Participants In Per-Protocol (PP) Analysis Set With Superficial and Deep Incisional SSI Involving Principal Incision Within 30 Days After the Index-surgery as Determined by Blinded Assessors 30 Days Post-operatively
Description: Superficial SSI: PD from SI, organisms isolated from aseptically obtained culture fluid from SI, pain/tenderness, localized swelling, redness, or heat extending from PI, or PI deliberately opened by surgeon for presumptive PI infection and was culture-positive, a negative wound culture but clinical evidence of infection on CIWS. Deep incisional SSI: PD from DI but not from organ/space component of the surgical site, fever (>38°C), localized wound pain, or wound tenderness, or DI spontaneously dehisces and/or deliberately opened by surgeon, and microbiological culture of DI by aseptic collection or deep wound swab was positive, an abscess or other evidence of infection involving DI was found on direct examination, during reoperation, or by histopathological or radiological examination, negative deep wound culture but clinical evidence of deep wound infection on CIWS.
Time Frame: Surgery (Day 0) up to 30 days post-surgery
Population: PP Analysis Set included all participants from ITT Analysis Set without any major protocol violations. Cumulative Treatment Incisional SSI was reported which included Superficial SSI and Deep SSI.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 197 | 196
Participants | 41 | 34
Statistical Analysis 1: Comparison: E-101 Solution 300 GU/mL vs Placebo (Saline Solution); Test type: Superiority; p = 0.34, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Clinical Infection Wound Scale Score (CIWS)
Description: CIWS was used postoperatively to evaluate the primary incisional wound for clinical evidence of infection. Score ranged from 0 (normal) - 5 (worst). 0: normal post-operative wound appearance, 1: wound erythema with pain extending ≥ 2 cm away from the primary incision, 2: spontaneous wound dehiscence with erythema and/or pain extending < 2 cm along primary incision, 3: spontaneous wound dehiscence with erythema and/or pain extending ≥ 2 cm along primary incision, 4: PD from the primary incision, 5: infection of primary incision involving deep incisional structures (muscle and/or fascia) manifested by one or more of the following: spontaneous partial or complete wound dehiscence with erythema and/or pain, spontaneous PD, a wound abscess (based on palpitation findings of the surgeon and/or needle aspiration of purulence into palpable fluctuance, and/or ultrasound examination above the fascia), clinical or histological evidence of fasciitis or myonecrosis.
Time Frame: Surgery (Day 0) up to 30 days post-surgery
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 235 | 220
score on a scale | 0.4 (1.09) | 0.4 (1.17)

4. Secondary Outcome: Number of Participants With Objectively Determined Incisional Surgical Site Infections (SSI)
Description: Number of participants with objectively determined SSI (defined as participants with PD, wound abscess, or positive microbial culture from one or more incisional samples) are reported.
Time Frame: Surgery (Day 0) up to 30 days post-surgery
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 241 | 225
Participants | 33 | 26

5. Secondary Outcome: Number of Participants With Superficial and Deep Incisional Surgical Site Infections (SSI) Involving the Principal Incision (PI) Within 30 Days After the Index-surgery as Determined by Blinded Assessors 14 Days Post-operatively
Description: Superficial SSI: PD from SI, organisms isolated from aseptically obtained culture fluid from SI, pain/tenderness, localized swelling, redness, or heat extending from PI, or PI deliberately opened by surgeon for presumptive PI infection and was culture-positive, a negative wound culture but CIWS. Deep incisional SSI: PD from DI but not from organ/space component of the surgical site, fever (>38°C), localized wound pain, or wound tenderness, or DI spontaneously dehisces and/or deliberately opened by a surgeon, and microbiological culture of DI by aseptic collection or deep wound swab was positive, an abscess or other evidence of infection involving DI was found on direct examination, during reoperation, or by histopathological or radiological examination, negative deep wound culture but clinical evidence of deep wound infection on CIWS.
Time Frame: Surgery (Day 0) up to 14 days post-surgery
Population: Participants in the ITT Analysis Set were analyzed. Cumulative Treatment Incisional SSI was reported which included Superficial SSI and Deep SSI.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 241 | 225
Participants | 50 | 52

6. Secondary Outcome: Worst Post-Baseline Mobility Score Using European Quality of Life-5 Dimensions (EQ-5D) Questionnaire
Description: The EQ-5D is a participant-answered questionnaire scoring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The mobility score questionnaire asked the participants to rate if they had problems walking around on a scale of 1 to 3 where 1= no problems, 2= some problems and 3= extreme problems. The mean worst post-baseline mobility scale score was presented.
Time Frame: Day 0 up to Day 30
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 190 | 178
score on a scale | 1.5 (0.56) | 1.6 (0.62)

7. Secondary Outcome: Worst Post-Baseline Self-Care Score Using European Quality of Life-5 Dimensions (EQ-5D) Questionnaire
Description: The EQ-5D is a participant-answered questionnaire scoring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The self-care questionnaire asked the participants to rate if they had any problems with self-care on a scale of 1 to 3 where 1= no problems, 2= some problems and 3= extreme problems. The mean worst post-baseline self-care scale score was presented.
Time Frame: Day 0 up to Day 30
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 190 | 178
score on a scale | 1.6 (0.68) | 1.6 (0.65)

8. Secondary Outcome: Worst Post-Baseline Usual Activity Score Using European Quality of Life-5 Dimensions (EQ-5D) Questionnaire
Description: The EQ-5D is a participant-answered questionnaire scoring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The usual activity questionnaire asked the participants to rate if they had any problems with usual activities on a scale of 1 to 3 where 1= no problems, 2= some problems and 3= extreme problems. The mean worst post-baseline usual activity scale score was presented.
Time Frame: Day 0 up to Day 30
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 190 | 178
score on a scale | 2.1 (0.64) | 2.0 (0.67)

9. Secondary Outcome: Worst Post-Baseline Pain/Discomfort Using European Quality of Life-5 Dimensions (EQ-5D) Questionnaire
Description: The EQ-5D is a participant-answered questionnaire scoring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The pain/discomfort score questionnaire asked the participants to rate if they had any pain or discomfort on a scale of 1 to 3 where 1= no problems, 2= some problems and 3= extreme problems. The mean worst post-baseline pain/discomfort scale score was presented.
Time Frame: Day 0 up to Day 30
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 190 | 178
score on a scale | 1.9 (0.53) | 1.9 (0.54)

10. Secondary Outcome: Worst Post-Baseline Anxiety/Depression Score Using European Quality of Life-5 Dimensions (EQ-5D) Questionnaire
Description: The EQ-5D is a participant-answered questionnaire scoring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The anxiety/depression questionnaire asked the participants to rate if they had any anxiety or depression on a scale of 1 to 3 where 1= no problems, 2= some problems and 3= extreme problems. The mean worst post-baseline anxiety/depression scale score was presented.
Time Frame: Day 0 up to Day 30
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 190 | 178
score on a scale | 1.4 (0.55) | 1.4 (0.60)

11. Secondary Outcome: Worst Post-Baseline Health State Score Using European Quality of Life-5 Dimensions (EQ-5D) Questionnaire
Description: The EQ-5D health state scale is a visual analog scale that ranges from 0 (worst imaginable health state) to 100 (best imaginable health state), with higher scores indicating a better state of health. Participants were asked to rate their health state from 0 to 100. The mean worst post-baseline health state score was reported.
Time Frame: Day 0 up to Day 30
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 190 | 178
score on a scale | 64.7 (20.77) | 61.3 (24.31)

12. Secondary Outcome: Number of Participants With Re-Hospitalization
Description: Number of participants who had re-hospitalization for SSI were reported.
Time Frame: Surgery (Day 0) up to 30 days post-surgery
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 241 | 225
Participants | 6 | 3

13. Secondary Outcome: Number of Participants With Clinical Wound Healing Score (CWHS) as Assessed by Blinded Assessors
Description: CWHS was assessed by blind assessors as 0= normal, intact incision without any spontaneous wound dehiscence; 1= spontaneous wound dehiscence that extends < 2 cm along the principal incision in the absence of erythema and/or pain 2= spontaneous wound dehiscence that extends ≥ 2 cm along the principal incision in the absence of erythema and/or pain. Number of participants with various levels of CWHS scores were reported.
Time Frame: Day 3 up to Day 30
Population: Participants in the Safety Analysis Set (all participants randomized to treatment and exposed to any quantity of study drug) with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 206 | 198
Participants
  CWHS =0 | 193 | 185
  CWHS =1 | 10 | 12
  CWHS =2 | 3 | 1

14. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-Emergent Adverse Events (TEAEs), Adverse Drug Reactions (ADRs), Suspected Unexpected Serious Adverse Reactions (SUSARs) and Unexpected Adverse Reactions (UARs)
Description: AE: Any untoward medical occurrence in a participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. ADR: All noxious and unintended responses to a medicinal product related to any dose. SAE: AE that resulted in any of the following: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE: an event that was not present prior to administration of study medication, or, if present prior to administration of study medication, increases in intensity after administration of study medication during study. SUSAR: all suspected adverse reactions (ARs) related to an investigational medicinal product (IMP) that occurred in study, and that were both unexpected and serious. UAR: an ARs, nature and severity of which was not consistent with the current medicinal product information.
Time Frame: From first dose up to 30 days post-surgery
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 248 | 234
Participants
  AEs | 218 | 202
  SAEs | 57 | 56
  TEAEs | 215 | 201
  ADRs | 10 | 10
  SUSARs | 0 | 0
  UARs | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Findings
Description: Number of participants with clinically significant laboratory findings were reported. The clinical significance was decided by the investigator.
Time Frame: From first dose up to 30 days post-surgery
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 248 | 234
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Number of participants with clinically significant physical examination findings were reported. The clinical significance was decided by the investigator.
Time Frame: From first dose up to 30 days post-surgery
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 248 | 234
Participants | 0 | 0

17. Secondary Outcome: Number of Participants by Wound Pain Assessment Scores
Description: Number of participants with wound pain assessment scores were assessed on a categorical scale ranging from 0 to 10, where 0 is no pain and 10 is unimaginable, unspeakable pain. Higher number on the scale represents worst possible pain.
Time Frame: Surgery (Day 0) up to 30 days post-surgery
Population: Participants in the Safety Analysis Set with available date were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 207 | 200
Participants
  Wound Pain Scale Score 0 | 8 | 9
  Wound Pain Scale Score 1 | 7 | 10
  Wound Pain Scale Score 2 | 15 | 20
  Wound Pain Scale Score 3 | 25 | 25
  Wound Pain Scale Score 4 | 37 | 26
  Wound Pain Scale Score 5 | 26 | 31
  Wound Pain Scale Score 6 | 29 | 26
  Wound Pain Scale Score 7 | 24 | 23
  Wound Pain Scale Score 8 | 23 | 18
  Wound Pain Scale Score 9 | 3 | 8
  Wound Pain Scale Score 10 | 10 | 4

18. Secondary Outcome: Number of Participants With pANCA Immunoglobulin G (IgG) Antibody, Serum Anti-glucose Oxidase (GO) IgG,M,A, pMPO IgG,M,A, Serum GO Neutralization, Serum pMPO Neutralization Antibody
Description: Antibody assessment was done using enzyme-linked immunosorbent assay (ELISA) test.
Time Frame: Day 14 and Day 30
Population: Participants in the Antibody Safety Set (all participants who were randomized to and exposed to any quantity of study drug with sufficient data to determine antibody results) with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 229 | 201
Participants
  pANCA IgG: Day 14: number analyzed (Participants) | 205 | 197
  pANCA IgG: Day 14 | 1 | 1
  pANCA IgG: Day 30 | 1 | 1
  Serum Anti-GO IgG,M,A: Day 14: number analyzed (Participants) | 204 | 197
  Serum Anti-GO IgG,M,A: Day 14 | 14 | 1
  Serum Anti-GO IgG,M,A: Day 30: number analyzed (Participants) | 220 | 200
  Serum Anti-GO IgG,M,A: Day 30 | 25 | 8
  Anti-pMPO IgG,M,A: Day 14: number analyzed (Participants) | 205 | 197
  Anti-pMPO IgG,M,A: Day 14 | 48 | 1
  Anti-pMPO IgG,M,A: Day 30: number analyzed (Participants) | 219 | 200
  Anti-pMPO IgG,M,A: Day 30 | 175 | 1
  Serum GO Neutralization: Day 14: number analyzed (Participants) | 13 | 1
  Serum GO Neutralization: Day 14 | 3 | 0
  Serum GO Neutralization: Day 30: number analyzed (Participants) | 23 | 6
  Serum GO Neutralization: Day 30 | 6 | 0
  Serum pMPO Neutralization: Day 14: number analyzed (Participants) | 50 | 2
  Serum pMPO Neutralization: Day 14 | 1 | 0
  Serum pMPO Neutralization: Day 30: number analyzed (Participants) | 171 | 1
  Serum pMPO Neutralization: Day 30 | 18 | 0

19. Secondary Outcome: Number of Participants With pANCA IgG Anti-body, Serum Anti-GO IgG,M,A, pMPO IgG,M,A, Serum Neutralization GO, Serum pMPO Neutralization Antibody
Description: Antibody assessment was done using ELISA test.
Time Frame: Month 3 and Month 6
Population: Participants in the Antibody Safety Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 71 | 2
Participants
  pANCA IgG: Month 3 | 0 | 0
  pANCA IgG: Month 6: number analyzed (Participants) | 32 | 0
  pANCA IgG: Month 6 | 0 |
  Serum Anti-GO IgG,M,A: Month 3: number analyzed (Participants) | 15 | 2
  Serum Anti-GO IgG,M,A: Month 3 | 3 | 1
  Serum Anti-GO IgG,M,A: Month 6: number analyzed (Participants) | 1 | 0
  Serum Anti-GO IgG,M,A: Month 6 | 1 |
  Anti-pMPO IgG,M,A: Month 3: number analyzed (Participants) | 70 | 1
  Anti-pMPO IgG,M,A: Month 3 | 60 | 0
  Anti-pMPO IgG,M,A: Month 6: number analyzed (Participants) | 33 | 0
  Anti-pMPO IgG,M,A: Month 6 | 31 |
  Serum GO Neutralization: Month 3: number analyzed (Participants) | 3 | 1
  Serum GO Neutralization: Month 3 | 0 | 0
  Serum GO Neutralization: Month 6: number analyzed (Participants) | 2 | 0
  Serum GO Neutralization: Month 6 | 0 |
  Serum pMPO Neutralization: Month 3: number analyzed (Participants) | 59 | 0
  Serum pMPO Neutralization: Month 3 | 14 |
  Serum pMPO Neutralization: Month 6: number analyzed (Participants) | 29 | 0
  Serum pMPO Neutralization: Month 6 | 5 |

20. Secondary Outcome: Number of Participants With Serum pANCA and pMPO Antibody Response
Time Frame: Day 30, Month 3 and Month 6
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
Number analyzed (Participants) | 248 | 234
Participants
  pANCA: Day 30 | 1 | 1
  pANCA: Month 3 | 0 | 0
  pANCA: Month 6 | 0 | 0
  Serum pMPO: Day 30 | 18 | 0
  Serum pMPO: Month 3 | 14 | 0
  Serum pMPO: Month 6 | 5 | 0

21. Other Pre Specified Outcome: Minimum Inhibitory Concentration (MIC) at 90%
Description: In vitro activity of the study drug against a range of aerobic and anaerobic pathogenic isolates cultured from infected principal incisions was analyzed using MIC. MIC 90 is defined as the lowest concentration of study drug that inhibits the growth of 90% of aerobic microorganisms tested.
Time Frame: Surgery (Day 0) up to to 30 days post surgery
Population: Per Protocol Analysis Set; only participant samples with isolated pathogens were included in the analysis
Measure: Number; unit: mg pMPO/mL
Units Other Than Participants: isolates
Arm/Group | E-101 Solution 300 GU/mL
Number analyzed (Participants) | 50
Number analyzed (isolates) | 76
mg pMPO/mL
  Aerobic | 0.25
  Anaerobic | NA — A lower threshold was not established (that is, the lowest possible administered doses inhibited anaerobic pathogens)

22. Other Pre Specified Outcome: Minimum Bactericidal Concentration (MBC) at 90%
Description: In vitro activity of the study drug against a range of aerobic and anaerobic pathogenic isolates cultured from infected principal incisions was analyzed using MBC. MBC 90 is defined as the lowest concentration of study drug required to kill greater than or equal to 99.9% (bactericidal) of the aerobic microorganisms tested.
Time Frame: Surgery (Day 0) up to to 30 days post surgery
Population: Per Protocol Analysis Set; only participant samples with isolated pathogens were included in the analysis
Measure: Number; unit: mg pMPO/mL
Units Other Than Participants: isolates
Arm/Group | E-101 Solution 300 GU/mL
Number analyzed (Participants) | 50
Number analyzed (isolates) | 76
mg pMPO/mL
  Aerobic | 0.5
  Anaerobic | NA — A lower threshold was not established (that is, the lowest possible administered doses inhibited anaerobic pathogens)

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days post-surgery
Description: Safety Analysis Set included all participants randomized to treatment and exposed to any quantity of study drug.
Arm/Group | E-101 Solution 300 GU/mL | Placebo (Saline Solution)
All-Cause Mortality (participants affected / at risk) | 2/248 | 2/234
Serious Adverse Events (participants affected / at risk) | 57/248 | 56/234
Other Adverse Events (participants affected / at risk) | 180/248 | 174/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E-101 Solution 300 GU/mL (N=248) | Placebo (Saline Solution) (N=234)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Diabetes insipidus (Endocrine disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 3 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2
Fat necrosis (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Secretion discharge (General disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 2 | 3
Abdominal infection (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 1 | 0
Pelvic infection (Infections and infestations) | 1 | 1
Pericolic abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 5
Post procedural sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 2
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Thrombophlebitis septic (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 7 | 9
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 2 | 4
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Ureteric injury (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abscess drainage (Surgical and medical procedures) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E-101 Solution 300 GU/mL (N=248) | Placebo (Saline Solution) (N=234)
Tachycardia (Cardiac disorders) | 27 | 29
Abdominal distension (Gastrointestinal disorders) | 20 | 28
Constipation (Gastrointestinal disorders) | 17 | 14
Diarrhoea (Gastrointestinal disorders) | 14 | 14
Dyspepsia (Gastrointestinal disorders) | 15 | 11
Nausea (Gastrointestinal disorders) | 98 | 93
Vomiting (Gastrointestinal disorders) | 34 | 40
Pyrexia (General disorders) | 38 | 35
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 13 | 8
Blood magnesium decreased (Investigations) | 11 | 18
Blood phosphorus decreased (Investigations) | 12 | 19
Haemoglobin decreased (Investigations) | 12 | 19
Oxygen saturation decreased (Investigations) | 13 | 17
Urine output decreased (Investigations) | 5 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 31 | 30
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 | 24
Hypophosphataemia (Metabolism and nutrition disorders) | 19 | 11
Insomnia (Psychiatric disorders) | 17 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 16
Hypotension (Vascular disorders) | 22 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No